CLINICAL TRIAL: NCT03313648
Title: A RCT Study of Laparoscopic Hepatectomy Versus RFA in the Treatment of Recurrent HCC
Brief Title: A Study of Laparoscopic Hepatectomy Versus RFA in the Treatment of Recurrent HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Institute of Hepatobiliary Surgery, Southwest Hospital, Third Military Medical University, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWHZSG007
Record Dates: First submitted 2017-10-05; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Hepatocellular Carcinoma Recurrent
Keywords: Recurrent HCC; Laparoscopic Hepatectomy; RFA; RCT
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Two different treatments are conducted on the participant base on the randomized choices
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Hepatectomy (Experimental): Improvements in laparoscopic technology mean that LH now has superior short-term efficacy and similar long-term efficacy to open surgery , and LH has shown significant advantages in applications involving recurrent HCC.
  Interventions: Procedure: Laparoscopic Hepatectomy
- Radiofrequency Ablation (Active Comparator): With recent technological advances, RFA has become the most widely investigated new first-line therapeutic option for recurrent HCCs . Numerous large studies have demonstrated the advantages of RFA, which include its ease of use, safety, effectiveness, minimal invasiveness, and minimal morbidity and mortality .
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Laparoscopic Hepatectomy — 180 patients with recurrent HCC with recurrent nodular diameters of less than 5 cm and up to three nodules were randomly divided into LH (n=90) and RFA groups (n=90). Outcomes were monitored and evaluated during the 5-year follow-up period.
  Arms: Laparoscopic Hepatectomy
Procedure: Radiofrequency Ablation — 180 patients with recurrent HCC with recurrent nodular diameters of less than 5 cm and up to three nodules were randomly divided into LH (n=90) and RFA groups (n=90). Outcomes were monitored and evaluated during the 5-year follow-up period.
  Arms: Radiofrequency Ablation

SUMMARY:
To observe and compare the short-term and long-term oncological outcome of laparoscopic hepatectomy and radiofrequency ablation in the treatment of recurrent hepatocellular carcinoma .

DETAILED DESCRIPTION:
Background & Aims: Hepatocellular carcinoma (HCC) is the third leading cause of cancer-related death in the world. The 5-year recurrent rate of HCC after first curative resection is 77%~100%. Laparoscopic repeat liver resection (LRLR) has been shown in small retrospective studies to be a safe and effective treatment for recurrent hepatocellular carcinoma (rHCC) in selected patients, and radiofrequency ablation (RFA) has been increasingly performed for treating recurrent tumors involving the liver after hepatectomy. The aim of this study was to compare the short-term and long-term outcome of laparoscopic hepatectomy (LH) and radiofrequency ablation (RFA) in the treatment of rHCC.

ELIGIBILITY:
Inclusion Criteria:

* Any gender,18 to 70 years old;
* Preoperative diagnosis of recurrent HCC clear,liver resection was done previously;
* No active hepatitis and decompensated cirrhosis;
* Patient with previous liver resection, maximum diameter ≤5cm single recurrent nodules or 3 nodules in diameter and no more than 3cm,did not infringe the portal vein,hepatic vein and inferior vena cava invasion,lymph node or extrahepatic turn;
* No tumor rupture or bleeding;
* Child-Pugh class A or B grade,ICG-R15 <20%;
* No coagulation disorders,platelet count > 50 × 109 / L and prolonged prothrombin time < 5 seconds;
* After diagnosis of recurrent HCC,not be including related surgery,radiofrequency ablation (RFA),TACE treatment,no certainty anticancer chemotherapy treatment;supreme absolute contraindications abdominal surgery;
* Recurrent nodules are not close to intestines,stomach,cholecyst or diaphragm muscle, not close to the first porta hepatis,main vessel and biliary ducts;
* Patients generally available,heart and lung function can tolerate surgery, abdominal surgery supreme absolute contraindications;
* Voluntarily participate in the study, voluntarily accept any therapy of two,informed consent.

Exclusion Criteria:

* Opposite of the above inclusion criteria;
* Severe upper abdominal adhesions;
* Postoperative pathological examination of the bile duct cell or mixed cell carcinoma and pathologically confirmed positive margin;
* Foreign,Hong Kong,Macao,Taiwan and other regions,estimated postoperative difficult to track,followed up;
* Nodules proved to be not recurrent HCC during intraoperative exploration, such as:liver metastases of colorectal cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 5 years
  follow-up after the surgery every 3 months, to understand statistics 5-year survival.

SECONDARY OUTCOMES:
intraoperative parameters | during the operation
  operation time and hepatic inflow occlusion time will be combined to report intraoperative parameters in hour(h).

OTHER OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  hepatic failure,hemorrhage,biliary leakage,ascites,intra-abdominal infection,pleural effusion,pulmonary infection,cardiac insufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China